CLINICAL TRIAL: NCT01804491
Title: Motion Analysis in Patients With Hallux Rigidus Before and After Different Types of Surgery
Brief Title: Motion Analysis in Patients With Hallux Rigidus
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. med. Benita Kuni, MD, Orthopedic and Trauma Surgeon, University Hospital Heidelberg
Other Study IDs: 252-2006-130228
Record Dates: First submitted 2013-03-01; First posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Hallux Rigidus
MeSH Terms: conditions — Hallux Rigidus

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Control group: Healthy age matched control subjects
  Interventions: Other: Motion Analysis
- Cheilectomy prospective group: Patients with hallux rigidus treated by the surgery type "cheilectomy"
  Interventions: Other: Motion Analysis
- Arthrodesis prospective group: Patients with hallux rigidus treated by the type of surgery "arthrodesis"
  Interventions: Other: Motion Analysis
- Mixed prospective group: Patients with hallux rigidus treated by other type of surgery: Arthoplasty, joint resection ("Keller-Brandes technique)
  Interventions: Other: Motion Analysis
- Cheilectomy retrospective group: Patients after cheilectomy due to hallux rigidus
  Interventions: Other: Motion Analysis
- Arthrodesis retrospective group: Patients after arthrodesis of the metatarsophalageal joint due to hallux rigidus
  Interventions: Other: Motion Analysis
- Mixed retrospective group: Patients after other types of surgery due to hallux rigidus: arthroplasty or resection of the first metatarso-phalangeal joint
  Interventions: Other: Motion Analysis

INTERVENTIONS:
Other: Motion Analysis — 3D Motion analysis with retroflective markers on the skin (Vicon camera system) of the foot and lower leg (kinematics), walking over force plate (kinetics) and pressure plates (plantar pressure distribution).

SUMMARY:
The aim was to investigate with a multi-segmental foot model the kinetic and kinematic in patients with a hallux rigidus, before and after different type of surgery.

DETAILED DESCRIPTION:
None of the patients received surgery BECAUSE of the study. We have only performed motion analysis in patients, who were already scheduled for one of the described type of surgery (prospective group) or who already previously received one the type of surgery (retrospective group).

ELIGIBILITY:
Inclusion Criteria:

* patients with osteoarthritis of one or both first metatarso-phalangeal joints (hallux rigidus)
* patients after surgery due to osteoarthritis of one or both first metatarso-phalangeal joints (hallux rigidus)

Exclusion Criteria:

* previous operations on the foot and ankle
* rheumatic diseases
* relevant foot deformities other than hallux rigidus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with osteoarthritis in the first metatarso-phalangeal joint (hallux rigidus)
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2006-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Change of hallux range of motion | baseline (=1 day before surgery) and 1 y. after surgery for the prospective groups, more than one year after surgery for the retrospective groups

CONTACTS AND LOCATIONS:
Locations (1):
- Motion Analysis Laboratory of the Department of Orthopedics, Trauma Surgery and Spinal Cord Injury, University Hospital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Kuni B, Wolf SI, Zeifang F, Thomsen M. Foot kinematics in walking on a level surface and on stairs in patients with hallux rigidus before and after cheilectomy. J Foot Ankle Res. 2014 Feb 13;7(1):13. doi: 10.1186/1757-1146-7-13. PMID 24524773